CLINICAL TRIAL: NCT05862428
Title: Rectal Misoprostol in Women Undergoing Total Abdominal Hysterectomy for Intraoperative Blood Loss Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Savang Vadhana Memorial Hospital, Thailand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 001/2022
Record Dates: First submitted 2023-04-23; First posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Intraoperative Blood Loss

STUDY DESIGN:
Intervention Model Description: The participants were devided in two groups. The experimental group received rectal misoprostol before surgery and the control group not received the drug
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rectal misoprostol (Experimental): This group received misoprostol transrectally before surgery 1 hour
  Interventions: Drug: Rectal misoprostol
- Control group (No Intervention): This group not received any drugs before surgery

INTERVENTIONS:
Drug: Rectal misoprostol — This intervention group receive Misoprostol transrectally before undergoing total abdominal hysterectomy
  Arms: Rectal misoprostol

SUMMARY:
Comparing of the intraoperative blood loss between group rectal misoprostol group and control group

DETAILED DESCRIPTION:
This open-labeled randomized controlled trial was conducted at the Department of Obstetrics and Gynecology, Queen Savang Vadhana Memorial Hospital, Chonburi, Thailand, from February 2022 to September 2022, after approval of the Institution of Review Board of Queen Savang Vadhana Memorial Hospital (IRB No. 001/2565).

Fifty six (56) women with diagnosis of benign uterine disease who were scheduled to perform total abdominal hysterectomy with or without bilateral salpingo-oophorectomy between February 2022 to September 2022 at Queen Savang Vadhana Memorial Hospital were enrolled in this study.

The participants were randomly allocated into two groups, study and control group. The randomization list was kept in a sealed opaque envelope. Study group received two tablets of 200 mcg misoprostol; The drug was inserted rectally 1 hour before operation. Few drops of normal saline were used to dissolve tablets before insertion. Control group that did not receive the drug. The drug was administered by a nurse at Gynecologic ward. The primary outcome was intraoperative blood loss that recorded by measuring amount of blood on the surgical gauzes and swabs by standardized scales and another was recorded from blood in suction container. The secondary outcome was hemoglobin differentiation, rate of blood transfusion and adverse events of misoprostol usage.

ELIGIBILITY:
Inclusion Criteria:

Female undergoing total abdominal hysterectomy (elective case) with

* No history of bleeding tendency
* No history of anticoagulant drug used within 7 days before surgery
* No contraindications of Misoprostol drug used
* No history of allergic to misoprostol

Exclusion Criteria:

* Can not communicate with Thai language
* Malignancy case
* Emergency case

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2022-02-18 (Actual); Primary Completion 2022-09-26 (Actual); Study Completion 2022-09-26 (Actual)

PRIMARY OUTCOMES:
Intraoperative blood loss | 7 months
  The intraoperative blood loss was defined as the blood at starting with a cut in the skin until the suture is closed. Its quantity was measure from blood pads and was record in millilitres. One gram of the blood was 1 ml.

SECONDARY OUTCOMES:
hemoglobin difference | 7 months
  The comparison of hemoglobin between the two groups.
Blood transfusion | 7 months
  Number of the participants between two groups that receive the blood component during or after the operation
Number of participants that have side effects of misoprostol | 7 months
  The comparison of frequencies of side effects of misoprostol between the two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Yingdhanai Pannaraj, Chon Buri, Changwat Chon Buri, Thailand

IPD SHARING:
Plan to Share IPD: No